CLINICAL TRIAL: NCT00952913
Title: A Study to Examine The Potential Effect Of Lansoprazole On The Pharmacokinetics Of Bosutinib When Administered Concomitantly To Healthy Subjects
Brief Title: Study Evaluating The Potential Effect Of Lansoprazole On The Pharmacokinetics Of Bosutinib In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3160A4-1108; B1871002
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
MeSH Terms: interventions — bosutinib; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bosutinib
  Interventions: Drug: Bosutinib
- 2 (Experimental): bosutinib + lansoprazole
  Interventions: Drug: Bosutinib; Drug: Lansoprazole

INTERVENTIONS:
Drug: Bosutinib — 4 x 100-mg oral tablets, single dose
  Other Names: SKI-606
  Arms: 1
Drug: Bosutinib — 4 x 100-mg oral tablets, single dose
  Other Names: SKI-606
  Arms: 2
Drug: Lansoprazole — 2 x 30-mg oral tablets, single daily doses for 2 days
  Other Names: Prevacid
  Arms: 2

SUMMARY:
The purpose of this study is to see if there is an effect on the pharmacokinetics of bosutinib when administered with lansoprazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of nonchildbearing potential, between the ages of 18 to 50 years old.

Exclusion Criteria:

* Any cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics as measured by Cmax, AUC, tmax, t1/2 | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Miami, Florida, United States

REFERENCES:
- [Derived] Abbas R, Leister C, Sonnichsen D. A clinical study to examine the potential effect of lansoprazole on the pharmacokinetics of bosutinib when administered concomitantly to healthy subjects. Clin Drug Investig. 2013 Aug;33(8):589-95. doi: 10.1007/s40261-013-0103-z. PMID 23839484
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3160A4-1108&StudyName=Study%20Evaluating%20The%20Potential%20Effect%20Of%20Lansoprazole%20On%20The%20Pharmacokinetics%20Of%20Bosutinib%20In%20Healthy%20Subjects